CLINICAL TRIAL: NCT04083599
Title: A First-in-Human, Open-label, Dose-escalation Trial With Expansion Cohorts to Evaluate Safety and Anti-tumor Activity of GEN1042 in Subjects With Malignant Solid Tumors
Brief Title: GEN1042 Safety Trial and Anti-tumor Activity in Participants With Malignant Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genmab (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCT1042-01; 2018-003716-47 (EudraCT Number); IRAS ID: 263292 (Registry Identifier: UK Research Summaries Database); MOH_2023-07-31_012855 (Registry Identifier: Israel MyTrials); 2023-508526-10 (Other: EU Trial (CTIS) Number); RECF-005255 (Other: National Institute of Cancer France); Rg13-835_03.08.2023 (Other: AMDM Moldova); 2023-508526-10-00 (EU CTIS Number)
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Malignant Solid Tumor; Non-Small Cell Lung Cancer (NSCLC); Colorectal Cancer (CRC); Melanoma; Head and Neck Squamous Cell Carcinoma (HNSCC); Pancreatic Ductal Adenocarcinoma (PDAC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Melanoma; Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab; Cisplatin; Carboplatin; Fluorouracil; Gemcitabine; Taxes; Pemetrexed; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Monotherapy - Dose Escalation and Dose Expansion Parts (Experimental)
  Interventions: Biological: GEN1042
- Combination Therapy - Safety Run-in and Expansion Parts (Experimental)
  Interventions: Biological: GEN1042; Drug: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: 5-FU; Drug: Gemcitabine; Drug: Nab paclitaxel; Drug: Pemetrexed; Drug: Paclitaxel

INTERVENTIONS:
Biological: GEN1042 — Intravenous
Drug: Pembrolizumab — Intravenous
  Arms: Combination Therapy - Safety Run-in and Expansion Parts
Drug: Cisplatin — Intravenous
  Arms: Combination Therapy - Safety Run-in and Expansion Parts
Drug: Carboplatin — Intravenous
  Arms: Combination Therapy - Safety Run-in and Expansion Parts
Drug: 5-FU — Intravenous
  Arms: Combination Therapy - Safety Run-in and Expansion Parts
Drug: Gemcitabine — Intravenous
  Arms: Combination Therapy - Safety Run-in and Expansion Parts
Drug: Nab paclitaxel — Intravenous
  Arms: Combination Therapy - Safety Run-in and Expansion Parts
Drug: Pemetrexed — Intravenous
  Arms: Combination Therapy - Safety Run-in and Expansion Parts
Drug: Paclitaxel — Intravenous
  Arms: Combination Therapy - Safety Run-in and Expansion Parts

SUMMARY:
The goal of this trial is to learn about the antibody GEN1042 when it is used alone and when it is used together with another antibody cancer drug, pembrolizumab (with or without chemotherapy), for treatment of participants with certain types of cancer.

DETAILED DESCRIPTION:
This is an open-label, multicenter phase 1/2 study designed to assess the safety, pharmacokinetics, pharmacodynamics and anti-tumor activity of GEN1042 administered as a monotherapy or in combination in participants with metastatic or locally advanced solid tumors.

Participants will receive either GEN1042 alone, GEN1042 with pembrolizumab, or GEN1042 with pembrolizumab and chemotherapy. All participants will receive active drug; no one will receive placebo.

This trial has 2 parts. The purpose of the first part is to find out if GEN1042 is safe and to find out the best doses of GEN1042 to use. The purpose of the second part is to give GEN1042 to more participants to see how well the dose(s) of GEN1042 selected in the first part work against cancer with GEN1042 when given alone or in combination with pembrolizumab or in combination with pembrolizumab and chemotherapy.

Trial details include:

* The average trial duration will be about 3 years.
* The treatment duration will be up to 2 years (when GEN1042 is combined with pembrolizumab).
* The visit frequency will be weekly at first and lessening over time until visits are only once every 3 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

Monotherapy - Dose Escalation and Dose Expansion Parts

* Participants with non-CNS solid tumors that is metastatic or unresectable and for whom there is no available standard therapy.
* Participants with a confirmed diagnosis of relapsed or refractory, advanced and/or metastatic melanoma, NSCLC, or CRC and for whom there is no available standard therapy

Combination Therapy - Dose Expansion Part

* Participants with unresectable Stage III or Stage IV melanoma with no prior systemic anticancer therapy for unresectable or metastatic disease. Primary ocular or mucosal melanoma is excluded.
* Participants with Stage IV metastatic or recurrent NSCLC with no prior systemic anticancer therapy, no actionable mutation.
* Participants with recurrent or metastatic HNSCC with no prior systemic therapy administered in the recurrent or metastatic setting.
* Participants with confirmed metastatic PDAC with no previous radiotherapy, surgery, chemotherapy, or investigational therapy for the treatment of metastatic disease.

General (all phases):

* Must be age ≥ 18 years of age on the day of signing informed consent, or the legal age of consent in the jurisdiction in which the trial is taking place.
* Measurable disease according to RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) 0-1
* Normal or adequate liver, renal, cardiac and bone marrow function

Key Exclusion Criteria:

Monotherapy - Dose Escalation and Dose Expansion Parts

* Treatment with an anti-cancer agent (within 21 days or after at least 5 half-lives of the drug, whichever is shorter), prior to GEN1042 administration
* Radiotherapy within 14 days prior to first GEN1042 administration
* Toxicities from previous anti-cancer therapies that have not resolved

Combination Therapy - Dose Expansion Part

* Has received prior systemic cytotoxic chemotherapy, biological therapy, OR major surgery within 3 weeks or at least 5 half-lives of the drug (whichever is shorter) of the first dose of trial treatment.
* Radiotherapy within 14 days of start of trial treatment or received lung radiation therapy of > 30 Gy within 6 months of the first dose of trial treatment.

General (all phases)

* Participants has an active, known, or suspected autoimmune disease.
* History of non-infectious pneumonitis that required steroids or currently has pneumonitis.
* History of ≥ grade 3 allergic reactions to monoclonal antibody (mAb) therapy
* Participants with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of first treatment.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation and Safety Run-in Parts: Number of Participants With Dose-Limiting Toxicities (DLTs) | First Cycle (21 days)
  Toxicities will be graded for severity according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) criteria version 5.0
Dose Expansion: Objective Response Rate (ORR) | Up to approximately 3 years
  ORR is defined as the percentage of participants with best overall response (BOR) [complete or partial response (PR or CR)] based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 as assessed by the investigator.

SECONDARY OUTCOMES:
All Parts: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From first dose until the end of the study (approximately 3 years)
Dose Escalation: ORR | Up to approximately 3 years
  ORR is defined as the percentage of participants with BOR (PR or CR) based on RECIST version 1.1 as assessed by the investigator.
All Parts: Duration of Objective Response (DOR) | Up to approximately 3 years
  DOR is defined as time from the first documentation of objective tumor response (CR or PR) to the date of first progressive disease (PD) or death based on RECIST version 1.1 as assessed by the investigator.
All Parts: Disease Control Rate (DCR) | Up to approximately 3 years
  DCR is defined as the percentage of participants with BOR of CR, PR, or stable disease (SD) based on RECIST version 1.1 as assessed by the investigator.
All Parts: Progression-Free Survival (PFS) | Up to approximately 3 years
  PFS is defined as the time from Day 1 in Cycle 1 to the first documented progression or death due to any cause based on RECIST version 1.1 as assessed by the investigator.
All Parts: Overall Survival (OS) | Up to approximately 3 years
  OS is defined as time from Day 1 in Cycle 1 to death due to any cause.
All Parts: Area Under the Concentration-Time Curve (AUC) of GEN1042 | Predose and postdose at multiple timepoints up to end of treatment (approximately 2 years)
All Parts: Maximum Observed Plasma Concentration (Cmax) of GEN1042 | Predose and postdose at multiple timepoints up to end of treatment (approximately 2 years)
All Parts: Half-life (t½) of GEN1042 | Predose and postdose at multiple timepoints up to end of treatment (approximately 2 years)
All Parts: Number of Participants With Anti-drug Antibody (ADA) Response to GEN1042 | Predose and postdose at multiple timepoints up to end of treatment (approximately 2 years)
  Serum samples will be screened for antibodies binding to GEN1042 and the titer of confirmed positive samples will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Genmab
Locations (76):
- United States (23):
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Cancer & Blood Specialty Clinic, Los Alamitos, California
  - Moores Cancer Center at the UC San Diego Health, San Diego, California
  - Yale University Cancer Center, New Haven, Connecticut
  - ChristianaCare, Newark, Delaware
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Florida Cancer Affiliates, Ocala, Florida
  - Hope and Healing Cancer Services, Hinsdale, Illinois
  - University of Kentucky, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Maryland Oncology Hematology PA, Columbia, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Levine Cancer Center, Charlotte, North Carolina
  - Novant Health Cancer Institute - Forsyth (Medical Oncology), Winston-Salem, North Carolina
  - Kaiser Permanente (KP) Oncology/Hematology, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Lumi Research, Kingwood, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Virgina Cancer Specialists, Fairfax, Virginia
  - Adventist Health System/Sunbelt,Inc, Seattle, Washington
  - Medical Oncology Associates, PS, Spokane, Washington
- Denmark (3):
  - Rigshospitalet (Copenhagen University Hospital), Copenhagen
  - Herlev University Hospital, Herlev
  - University Hospital of Southern Denmark, Vejle Hospital, Vejle
- France (3):
  - Centre hospitalier Universitaire de Bordeaux, Bordeaux
  - Centre Antoine Lacassagne, Nice
  - Gustave Roussy, Villejuif
- ARENSIA Research Clinic at the Research Institute of Clinical Medicine, Tbilisi, Georgia
- Germany (5):
  - Nationales Centrum fr Tumorerkrankungen NCT, Heidelberg
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen
  - Department of Dermatology, University of Mainz, Mainz
  - UniversitÃ¤tsmedizin Mannheim Dermatologie, Mannheim
  - Universitaetsklinikum Wuerzburg, Würzburg
- Israel (2):
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (4):
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera S.Croce e Carle Cuneo, Cuneo
  - Istituto Nazionale dei Tumori, Milan
  - Istituto Clinico Humanitas, Rozzano
- ARENSIA Research Clinic at the Oncology Institute, Chisinau, Moldova
- South Korea (7):
  - Chungbuk National University Hospital, Cheongju-si
  - Jeonbuk National University Hospital, Jeonju
  - Gachon University Gil Medical Center, Namdong
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Pusan National University Yangsan Hospital, Yangsan
- Spain (19):
  - H. Vall d'Hebron, Barcelona
  - START Barcelona HM Nou Delfos, Barcelona
  - Hospital Duran i Reynals - ICO L Hospitalet, L'Hospitalet de Llobregat
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Universitario Lucus Augusti, Lugo
  - Clinica Universidad de Navarra, Madrid
  - HM CIOCC Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital General Universitario Gregorio Maran, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - MD Anderson Cancer Center Madrid, Madrid
  - START Madrid - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Clinica Universidad de Navarra, Pamplona
  - Complejo Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela
  - Hospital Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- Taiwan (7):
  - Chang Gung Memorial Hospital (CGMH) - Kaohsiung Branch, Kaohsiung City
  - Kaohsiung Medical University Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, VGHTPE, Taipei
  - Chang Gung Memorial Hospital Linkou Branch, Taoyuan District
- Royal Marsden NHS Foundation Trust, Sutton, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muik A, Adams 3rd HC, Gieseke F, Altintas I, Schoedel KB, Blum JM, Sanger B, Burm SM, Stanganello E, Verzijl D, Spires VM, Vascotto F, Toker A, Quinkhardt J, Fereshteh M, Diken M, Satijn DPE, Kreiter S, Ahmadi T, Breij ECW, Tureci O, Sasser K, Sahin U, Jure-Kunkel M. DuoBody-CD40x4-1BB induces dendritic-cell maturation and enhances T-cell activation through conditional CD40 and 4-1BB agonist activity. J Immunother Cancer. 2022 Jun;10(6):e004322. doi: 10.1136/jitc-2021-004322. PMID 35688554